CLINICAL TRIAL: NCT00953212
Title: A Randomized Controlled Trial to Compare Prophylaxis With Oral Ascorbic Acid, Oral Amiodarone or Both in Combination With Beta Blockers to Reduce Postoperative Atrial Fibrillation After Cardiac Surgery
Brief Title: Prophylaxis to Reduce Postoperative Atrial Fibrillation in Cardiac Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MaineHealth (Other)
Responsible Party: Principal Investigator, Peter C. Donovan, Staff Physician Assistant, Cardiothoracic Surgery, MaineHealth
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: MMC-3514
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-03

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: atrial fibrillation; cardiac surgery; open heart surgery
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter | interventions — Adrenergic beta-Antagonists; Metoprolol; Amiodarone; Ascorbic Acid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A (Active Comparator): Beta Blockers, Ascorbic Acid and Amiodarone
  Interventions: Drug: beta blockers; Drug: amiodarone; Drug: ascorbic acid
- Group B (Active Comparator): Beta Blockers and Ascorbic Acid
  Interventions: Drug: beta blockers; Drug: ascorbic acid
- Group C (Active Comparator): Beta Blockers and Amiodarone
  Interventions: Drug: beta blockers; Drug: amiodarone
- Group D (Active Comparator): Beta Blockers alone
  Interventions: Drug: beta blockers

INTERVENTIONS:
Drug: beta blockers — metoprolol 25mg by mouth every 6 hours
  Other Names: Lopressor; Toprol XL
Drug: amiodarone — amiodarone 600mg by mouth evening before surgery amiodarone 600mg by mouth morning of surgery amiodarone 400mg by mouth every 12 hours for 3 days postoperatively
  Other Names: Cordarone
  Arms: Group A; Group C
Drug: ascorbic acid — ascorbic acid 2,000mg by mouth evening before surgery ascorbic acid 2,000mg by mouth morning of surgery ascorbic acid 1,000mg by mouth every 12 hours for 5 postoperative days
  Other Names: vitamin C
  Arms: Group A; Group B

SUMMARY:
Atrial Fibrillation (AF) is a common postoperative complication of cardiac surgery, occuring in approximately 25-30% of coronary artery bypass graft (CABG) patients and 35-40% of heart valve repair/replacement patients. Efforts to decrease the high rates of AF have not made great inroads to the problem. The current standard of care is the use of preoperative and postoperative beta blockers. We propose to compare the use of prophylactic oral ascorbic acid with and without prophylactic oral amiodarone, in combination with oral beta blockers, for the prevention of atrial fibrillation after open heart surgery. The hypothesis is that either drug, or a combination of the two drugs, will be superior and safe when compared to beta blockers alone.

DETAILED DESCRIPTION:
Atrial fibrillation is a common complication of cardiac surgery which is associated with increased morbidity, length of stay and cost. Efforts to mitigate this problem with beta blockers and amiodarone have been met with limited success. Observational data suggests that prophylactic amiodarone has been helpful in decreasing the incidence of AF as well as increasing its ease of management. The opportunity to use ascorbic acid for AF prophylaxis is attractive because of its low side effect profile, wide acceptance and low cost.

We have designed a prospective, randomized, controlled trial using a 2 X 2 factorial design to determine whether prophylactic ascorbic acid alone, ascorbic acid with amiodarone, or amiodarone alone, when given along with beta blockers will decrease the incidence of postoperative AF in adult cardiac surgery in all comers as compared with beta blockers alone.

Patients will be randomized into four groups, A, B, C, and D. All groups will receive beta blockers, Group A will receive beta blockers, ascorbic acid, and amiodarone, Group B will receive ascorbic acid and Beta blockers, Group C will receive amiodarone and beta blockers and Group D will receive only beta blockers.

Success of randomization will be assessed by comparing treatment groups with respect to baseline characteristics, using t-tests or their nonparametric equivalent (as appropriate) for continuous variables and chisquare tests or Fisher's exact tests for categorical variables. The primary hypotheses of the effects of ascorbic acid and amiodarone on incidence of atrial fibrillation will be tested using chisquare tests for differences in proportions. No adjustment will be made for multiple comparisons since both hypotheses are pre-specified. We will use exploratory analyses including stratification to assess for the possibility of effect modification between ascorbic acid and amiodarone. If an interaction is suggested by these analyses, we will use logistic regression with a cross-product term as a formal statistical test for interaction.

ELIGIBILITY:
Inclusion Criteria:

* adults (18 years of age or older)
* all comers for elective or urgent open heart surgery ( CABG, Valve repair or replacement, Combined CABG/Valves, CABG/other, Other)

Exclusion Criteria:

* patients who refuse to participate
* patients with a history of atrial fibrillation or atrial flutter
* pediatric patients (under 18 years of age)
* Emergency surgery
* patients with contraindications to study medications
* patients with untreated thyroid disease, hepatic failure, pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2009-08; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Donovan, PA-C, MHS, Principal Investigator — MaineHealth; Robert S Kramer, M.D., Study Chair — MaineHealth
Locations (1):
- Maine Medical Center, Portland, Maine, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Beta Blockers, Ascorbic Acid and Amiodarone: beta blockers: metoprolol 25mg by mouth every 6 hours
  amiodarone: amiodarone 600mg by mouth evening before surgery amiodarone 600mg by mouth morning of surgery amiodarone 400mg by mouth every 12 hours for 3 days postoperatively
  ascorbic acid: ascorbic acid 2,000mg by mouth evening before surgery ascorbic acid 2,000mg by mouth morning of surgery ascorbic acid 1,000mg by mouth every 12 hours for 5 postoperative days
- Beta Blockers and Ascorbic Acid: Beta Blockers and Ascorbic Acid beta blockers: metoprolol 25mg by mouth every 6 hours
  ascorbic acid: ascorbic acid 2,000mg by mouth evening before surgery ascorbic acid 2,000mg by mouth morning of surgery ascorbic acid 1,000mg by mouth every 12 hours for 5 postoperative days
- Beta Blockers and Amiodarone: Beta Blockers and Amiodarone
  beta blockers: metoprolol 25mg by mouth every 6 hours
  amiodarone: amiodarone 600mg by mouth evening before surgery amiodarone 600mg by mouth morning of surgery amiodarone 400mg by mouth every 12 hours for 3 days postoperatively
- Beta Blockers Alone: Beta Blockers alone
  beta blockers: metoprolol 25mg by mouth every 6 hours
Period: Overall Study
Arm/Group | Beta Blockers, Ascorbic Acid and Amiodarone | Beta Blockers and Ascorbic Acid | Beta Blockers and Amiodarone | Beta Blockers Alone
Started | 76 | 74 | 78 | 76
Completed | 76 | 74 | 78 | 76
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Group D | Total
Number analyzed (Participants) | 76 | 74 | 78 | 76 | 304
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (9.6) | 65.9 (9.4) | 63.9 (10.7) | 33.4 (931) | 61 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 19 | 20 | 74
  Male | 60 | 55 | 59 | 56 | 230
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 76 | 74 | 77 | 75 | 302
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Smoker [Count of Participants; unit: Participants] | 16 | 19 | 21 | 19 | 75
BMI (mean, SD) [Mean (Standard Deviation); unit: kg/m^2] | 30.6 (6.1) | 31.1 (5.7) | 27.9 (4.7) | 29.5 (6.2) | 29.7 (5.8)
Cardiovascular Disease [Count of Participants; unit: Participants] | 11 | 13 | 14 | 13 | 51
Hypertension [Count of Participants; unit: Participants] | 69 | 63 | 62 | 65 | 259
Pre-op Myocardial Infarction [Count of Participants; unit: Participants] | 24 | 30 | 29 | 35 | 118
Diabetes [Count of Participants; unit: Participants] | 28 | 28 | 23 | 27 | 106
Peripheral Vascular Disease [Count of Participants; unit: Participants] | 10 | 8 | 9 | 10 | 37
Chronic Obstructive Pulmonary Disease [Count of Participants; unit: Participants] | 10 | 7 | 3 | 11 | 31
Statin [Count of Participants; unit: Participants] | 54 | 50 | 52 | 47 | 203
Congestive Heart Failure [Count of Participants; unit: Participants] | 6 | 8 | 4 | 8 | 26
Surgery Type - CABG [Count of Participants; unit: Participants] | 62 | 57 | 55 | 58 | 232
Surgery Type - Valve [Count of Participants; unit: Participants] | 6 | 6 | 13 | 3 | 28
Surgery Type - CABG/Valve [Count of Participants; unit: Participants] | 6 | 9 | 9 | 12 | 36
Surgery Type - Other [Count of Participants; unit: Participants] — Other surgeries include ascending aortic repair, myxoma excision, patent ductus foramen ovale closure, or endarterectomy
  Participants | 2 | 2 | 1 | 3 | 8
Urgent Surgery [Count of Participants; unit: Participants] | 68 | 72 | 71 | 73 | 284

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Post-operative Atrial Fibrillation Requiring Treatment After Open Heart Surgery
Description: Atrial fibrillation is a common complication of cardiac surgery which is associated with increased morbidity, length of stay and cost. The opportunity to use ascorbic acid for AF prophylaxis is attractive because of its low side effect profile, wide acceptance and low cost. This prospective, randomized trial used a 2 X 2 factorial design to determine whether prophylactic ascorbic acid alone, ascorbic acid with amiodarone, or amiodarone alone, when given along with beta blockers would decrease the incidence of postoperative AF in adult cardiac surgery when compared with beta blockers alone, all combinations failed to show any difference between the four groups. While there have been trials that have shown the addition of amiodarone to beta-blockers to be more effective, this analysis does not support that conclusion.
Time Frame: 5 postoperative days
Population: Number of patients who experienced Atrial Fibrillation post-operatively
Measure: Count of Participants; unit: Participants
Groups:
- Amiodarone - Yes: Patients who were administered Amiodarone and Beta Blockers with or without Ascorbic Acid.
- Amiodarone - No: Patients who were not administered Amiodarone and Beta Blockers with or without Ascorbic Acid.
- Ascorbic Acid - Yes: Patients who were administered Ascorbic Acid and Beta Blockers with or without Amiodarone.
- Ascorbic Acid - No: Patients who were not administered Ascorbic Acid and Beta Blockers with or without Amiodarone.
Arm/Group | Amiodarone - Yes | Amiodarone - No | Ascorbic Acid - Yes | Ascorbic Acid - No
Number analyzed (Participants) | 154 | 150 | 150 | 154
Participants | 50 | 56 | 58 | 48

2. Secondary Outcome: Number of Participants With Mortality
Description: Mortality measured within length of hospital stay
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Beta Blockers, Ascorbic Acid and Amiodarone | Beta Blockers and Ascorbic Acid | Beta Blockers and Amiodarone | Beta Blockers Alone
Number analyzed (Participants) | 154 | 150 | 150 | 154
Participants | 1 | 1 | 1 | 0

3. Secondary Outcome: Hospital Length of Stay
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Amiodarone - Yes | Amiodarone - No | Ascorbic Acid - Yes | Ascorbic Acid - No
Number analyzed (Participants) | 154 | 150 | 150 | 154
days | 7.0 (4.8) | 6.6 (3.8) | 6.8 (3.6) | 6.8 (4.9)

4. Secondary Outcome: ICU Length of Stay
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Amiodarone - Yes | Amiodarone - No | Ascorbic Acid - Yes | Ascorbic Acid - No
Number analyzed (Participants) | 154 | 150 | 150 | 154
days | 2.0 (1.5) | 1.9 (1.3) | 2.0 (1.3) | 1.9 (1.5)

5. Secondary Outcome: Number of Participants With Stroke
Description: Cerebral vascular accident occurring within hospital length of stay
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Amiodarone - Yes | Amiodarone - No | Ascorbic Acid - Yes | Ascorbic Acid - No
Number analyzed (Participants) | 154 | 150 | 150 | 154
Participants | 1 | 3 | 1 | 1

6. Secondary Outcome: Number of Participants With Low Output Heart Failure
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Amiodarone - Yes | Amiodarone - No | Ascorbic Acid - Yes | Ascorbic Acid - No
Number analyzed (Participants) | 154 | 150 | 150 | 154
Participants | 12 | 10 | 7 | 9

7. Secondary Outcome: Number of Participants With Postoperative Vasoplegia
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Amiodarone - Yes | Amiodarone - No | Ascorbic Acid - Yes | Ascorbic Acid - No
Number analyzed (Participants) | 154 | 150 | 150 | 154
Participants | 17 | 15 | 14 | 16

8. Secondary Outcome: Number of Participants With Respiratory Failure Requiring Reintubation
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Amiodarone - Yes | Amiodarone - No | Ascorbic Acid - Yes | Ascorbic Acid - No
Number analyzed (Participants) | 154 | 150 | 150 | 154
Participants | 4 | 2 | 2 | 5

9. Secondary Outcome: Number of Participants With Bradycardia Necessitating Permanent Pacemaker Placement
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Amiodarone - Yes | Amiodarone - No | Ascorbic Acid - Yes | Ascorbic Acid - No
Number analyzed (Participants) | 154 | 150 | 150 | 154
Participants | 0 | 2 | 0 | 2

10. Secondary Outcome: Number of Participants With Acute Kidney Injury
Description: Using the Akin definition
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Amiodarone - Yes | Amiodarone - No | Ascorbic Acid - Yes | Ascorbic Acid - No
Number analyzed (Participants) | 154 | 150 | 150 | 154
Participants | 19 | 13 | 22 | 11

11. Secondary Outcome: Number of Participants With Readmission to ICU for Treatment of Atrial Fibrillation
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Amiodarone - Yes | Amiodarone - No | Ascorbic Acid - Yes | Ascorbic Acid - No
Number analyzed (Participants) | 154 | 150 | 150 | 154
Participants | 1 | 1 | 2 | 0

12. Secondary Outcome: Number of Participants With Readmission to Hospital for Treatment of Atrial Fibrillation
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Amiodarone - Yes | Amiodarone - No | Ascorbic Acid - Yes | Ascorbic Acid - No
Number analyzed (Participants) | 154 | 150 | 150 | 154
Participants | 4 | 4 | 4 | 4

ADVERSE EVENTS:
Arm/Group | Group A | Group B | Group C | Group D
All-Cause Mortality (participants affected / at risk) | 1/76 | 1/74 | 1/78 | 0/76
Serious Adverse Events (participants affected / at risk) | 1/76 | 3/74 | 1/78 | 1/76
Other Adverse Events (participants affected / at risk) | 29/76 | 29/74 | 21/78 | 27/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=76) | Group B (N=74) | Group C (N=78) | Group D (N=76)
Cerebral Vascular Accident (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=76) | Group B (N=74) | Group C (N=78) | Group D (N=76)
Atrial fibrillation (Cardiac disorders) | 29 (29) | 29 (29) | 21 (21) | 27 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes